CLINICAL TRIAL: NCT04895943
Title: Influence of Bariatric Endoscopy on Clinical Course of NAFLD
Brief Title: Bariatric Endoscopy and NAFLD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: 04_RVO-FNOs_2021
Record Dates: First submitted 2021-05-05; First posted 2021-05-21 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Obesity; NAFLD; Liver Steatosis; Liver Fibrosis
Keywords: Obesity; NAFLD; liver steatosis; liver fibrosis; bariatric endoscopy; weight loss
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Cirrhosis; Weight Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with adjustable IGB
  Interventions: Procedure: bariatric endoscopy, mainly intragastric balloons, plication of the stomach too
- Group with non-adjustable IGB
  Interventions: Procedure: bariatric endoscopy, mainly intragastric balloons, plication of the stomach too

INTERVENTIONS:
Procedure: bariatric endoscopy, mainly intragastric balloons, plication of the stomach too — bariatric endoscopy, mainly intragastric balloons, plication of the stomach too
  Groups: Group with adjustable IGB
Procedure: bariatric endoscopy, mainly intragastric balloons, plication of the stomach too — bariatric endoscopy, mainly intragastric balloons, plication of the stomach too
  Groups: Group with non-adjustable IGB

SUMMARY:
Find out how bariatric endoscopy will influence the clinical course of non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
The study will test and investigate the impact of bariatric endoscopy (various types of intragastric balloons, endoscopic sleeve gastroplasty, aspiration therapy) on components of the metabolic syndrome in obese patients, especially on influencing non-alcoholic steatosis and steatohepatitis and signs of liver fibrotization and weight reduction. The method consists of performing a mini-invasive endoscopic procedure and, as a result, reduced food intake.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21-70 years
* BMI >27 Kg/m2
* Must be able to comply with all study requirements for the duration of the study as outlined in the protocol. This includes complying with the visit schedule as well as study-specific procedures such as clinical assessment, endoscopy, radiography, as well as laboratory investigations
* Must be able to understand and be willing to provide written informed consent
* Patient living within radio range 300 km from the study center
* Failure of the cognitive-behavioral approach to weight reduction

Exclusion Criteria:

Subjects meeting any of the following exclusionary criteria cannot be enrolled in the study:

* BMI <27
* History of gastric surgery.
* Previous technical difficulties in gastric and duodenal endoscopy or inability to perform endoscopy
* History of GIT diseases such as achalasia, esophageal motility disorders, severe esophagitis or gastritis, the recent history of ulcers, history of steatosis or obstruction in the GIT
* Proven celiac disease
* Previous irreversible endoscopic procedures and surgical treatment of obesity
* Chronic and acute pancreatitis
* Active or chronic infectious hepatitis
* Known liver disease or suspected PBC, PSC, autoimmune hepatitis, alpha1-antitrypsin deficiency, Wilson's disease, hereditary hemochromatosis, known cirrhosis or history of hepatic decompensation, AST or ALT> 5-8x ULN
* Type 1 or type 2 diabetes with insulin
* History of malignant disease
* Specific genetic or hormonal disorders associated with obesity (Prader-Willi syndrome, MC4R mutations, etc.)
* Serious disorders of blood clotting and hematopoiesis
* Severe forms of psychiatric illness (endogenous depression, schizophrenia, suicidal tendencies, psychosis)
* Uncontrolled hypertension (systolic BP> 150 mm Hg or diastolic BP> 100 mm Hg) or severe heart disease (severe cardiac dysfunction, etc.)
* Serious autoimmune diseases or long-term use treated with glucocorticoids or immunosuppressive therapy
* Disorders of thyroid function unresponsive to processing.
* Renal impairment with GFR <60 ml / min / 1.73 m2, or albumin excretion> 1000 mg / day
* Substance use including excessive alcohol use (> 21 units / week for men and> 14 units / week for women, - 1 unit (250ml 12 ° or 330ml 10 ° beer; 100ml wine; 25ml = small spirits of spirits))
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients undergoing bariatric endoscopy procedure.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with NAFLD with degree of fibrosis of the liver among patients undergoing bariatric endoscopy and to determine the influence of bariatric endoscopy on clinical course of NAFLD and liver fibrosis | 24 months
  Number of patients with NAFLD with degree of fibrosis of the liver among patients undergoing bariatric endoscopy and to determine the influence of bariatric endoscopy on clinical course of NAFLD and liver fibrosis

SECONDARY OUTCOMES:
Influence of bariatric endoscopy on change of weight | 24 months
  Influence of bariatric endoscopy on change of weight
Influence of bariatric endoscopy on change of anthropometric parameters | 24 months
  Influence of bariatric endoscopy on change of anthropometric parameters
Anthropometric changes - weight (kg), BMI (kg/m2) | 24 months
  Anthropometric changes - weight (kg), BMI (kg/m2)
Anthropometric changes - waist and hip circumference (cm) | 24 months
  Anthropometric changes - waist and hip circumference (cm)
Nutritional changes (eating habits) - questionnaire survey. | 24 months
  Nutritional changes (eating habits) - questionnaire survey.
Components of the metabolic syndrome - blood pressure (mm/Hg) | 24 months
  Components of the metabolic syndrome - blood pressure (mm/Hg)
Components of the metabolic syndrome - waist circumference (cm) | 24 months
  Components of the metabolic syndrome - waist circumference (cm)
Components of the metabolic syndrome - triacylglycerol levels (mmol/l), HDL cholesterol levels (mmol/l), glycemia (mmol/l) | 24 months
  Components of the metabolic syndrome - triacylglycerol levels (mmol/l), HDL cholesterol levels (mmol/l), glycemia (mmol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Vašura, MD, Study Chair — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Fakhry TK, Mhaskar R, Schwitalla T, Muradova E, Gonzalvo JP, Murr MM. Bariatric surgery improves nonalcoholic fatty liver disease: a contemporary systematic review and meta-analysis. Surg Obes Relat Dis. 2019 Mar;15(3):502-511. doi: 10.1016/j.soard.2018.12.002. Epub 2018 Dec 6. PMID 30683512
- [Background] Machytka E, Klvana P, Kornbluth A, Peikin S, Mathus-Vliegen LE, Gostout C, Lopez-Nava G, Shikora S, Brooks J. Adjustable intragastric balloons: a 12-month pilot trial in endoscopic weight loss management. Obes Surg. 2011 Oct;21(10):1499-507. doi: 10.1007/s11695-011-0424-z. PMID 21553304
- [Background] Leoni S, Tovoli F, Napoli L, Serio I, Ferri S, Bolondi L. Current guidelines for the management of non-alcoholic fatty liver disease: A systematic review with comparative analysis. World J Gastroenterol. 2018 Aug 14;24(30):3361-3373. doi: 10.3748/wjg.v24.i30.3361. PMID 30122876
- [Derived] Vasura A, Machytka E, Urban O, Machackova J, Pavliska L, Berka Z, Svagera Z, Buzga M. Effect of bariatric endoscopy on liver fibrosis and steatosis and the course of NAFLD - a prospective interventional study. Ann Hepatol. 2025 Jan-Jun;30(1):101765. doi: 10.1016/j.aohep.2024.101765. Epub 2024 Dec 12. PMID 39674369